CLINICAL TRIAL: NCT00044057
Title: A Multicenter, Stratified, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate Neurologic Function and Disability in Patients With Acute Ischemic Stroke Given Tissue Plasminogen Activator Plus YM872 or Tissue Plasminogen Activator Plus Placebo
Brief Title: A Study to Evaluate the Effects of YM872 on Brain Function and Disability When Administered in Combination With Alteplase (Tissue Plasminogen Activator)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: Astellas Pharma US, Inc. (Industry)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: 872-CL-004
Record Dates: First submitted 2002-08-16; First posted 2002-08-20 (Estimated); Last update posted 2006-04-03 (Estimated); Status verified 2006-03

CONDITIONS: Acute Ischemic Stroke
Keywords: ARTIST
MeSH Terms: conditions — Ischemic Stroke | interventions — YM 872; Tissue Plasminogen Activator

INTERVENTIONS:
Drug: YM872 (zonampanel), t-PA (alteplase)

SUMMARY:
The purpose of this study is to determine if YM872 in combination with t-PA can reduce disability and brain damage from stroke. YM872 or placebo will be given as a continuous intravenous (iv) infusion for 24 hours. It is important that the study medication, YM872 or placebo, is administered prior to the completion of the t-PA administration. The clinical effects of YM872 in addition to t-PA will be determined by assessing neurological function and disability scores at follow up visits through Day 90 of the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute ischemic stroke who are treated with alteplase within 3 hours of stroke onset (Onset is defined as the time that which the patient was last seen in a normal state, or bedtime for unwitnessed strokes occurring during the night).
* Patients who are able to provide written informed consent or have consent provided by a legally authorized representative.
* Patients who are at least 18 years of age.
* Patients who have a National Institutes of Health Stroke Scale (NIHSS) score of at least 7 but not more than 23 and who are conscious.
* Other criteria as specified in the study protocol

Exclusion Criteria:

* Patients who are not eligible to receive treatment with alteplase (t-PA) due to brain hemorrhage, risk for hemorrhage, or other criteria.
* Patients who have stroke of the brainstem or cerebellum.
* Patients who have renal (kidney) disease or insufficiency.
* Patients who have active epilepsy or convulsions during the current stroke episode.
* Patients who are IV drug users or are inebriated.
* Patients who have a history of drug-related anaphylaxis.
* Patients who have taken sedatives, anticonvulsants, or any medication with sedating effects in the 10 days prior study enrollment.
* Patients who have taken more than 1.3 g of aspirin per day in the 2 days prior to enrollment.
* Patients who have a known vitamin hypersensitivity.
* Other exclusion criteria as specified by the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-12; Study Completion 2003-01

CONTACTS AND LOCATIONS:
Locations (118):
- United States (94):
  - University of South Alabama Stroke Center, Mobile, Alabama
  - Good Samaritan Hospital, Phoenix, Arizona
  - University of Arizona, Tucson, Arizona
  - East Bay Region Associates in Neurology, Berkeley, California
  - Providence St. Joseph's Medical Center, Burbank, California
  - Mercy San Juan Hospital, Carmichael, California
  - University of California Davis Medical Center, Davis, California
  - Scripps Memorial Hospital, Encinitas, California
  - Grossmont Hospital, La Mesa, California
  - UCLA Medical Center, Los Angeles, California
  - Tri-City Medical Center, Oceanside, California
  - Stanford University Medical Center, Palo Alto, California
  - Mercy General Hospital, Sacramento, California
  - Scripps Mercy Hospital, San Diego, California
  - University of California at San Diego, San Diego, California
  - Good Samaritan Hospital, San Jose, California
  - UCLA Medical Center - Santa Monica, Santa Monica, California
  - John Muir Medical Center, Walnut Creek, California
  - Mt Diablo Medical Center, Walnut Creek, California
  - Colorado Neurological Institute, Englewood, Colorado
  - Bridgeport Hospital, Bridgeport, Connecticut
  - Columbia JFK Hospital, Atlantis, Florida
  - Bethesda Memorial Hospital, Boynton Beach, Florida
  - Lakeland Regional Medical Center, Lakeland, Florida
  - Holmes Regional Medical Center, Melbourne, Florida
  - Bay Medical Center, Panama City, Florida
  - St Joseph's Hospital, Tampa, Florida
  - Tampa General Hospital, Tampa, Florida
  - St Francis Hospital, Columbus, Georgia
  - DNA Research (Dekalb Medical Center), Decatur, Georgia
  - Candler Hospital, Savannah, Georgia
  - St Joseph Hospital, Savannah, Georgia
  - Queen's Medical Center, Honolulu, Hawaii
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Parkview Hospital, Fort Wayne, Indiana
  - Methodist Hospital, Indianapolis, Indiana
  - Louisville Neuroscience Research Center, Louisville, Kentucky
  - Culicchia Neurology Clinic, LLP, Marrero, Louisiana
  - University of Maryland Medical System, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - New England Medical Center, Boston, Massachusetts
  - St John's Hospital, Detroit, Michigan
  - Michigan State University, East Lansing, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - Northern Michigan Neurology, Traverse City, Michigan
  - Bi-County Hospital, Warren, Michigan
  - Research Medical Center, Kansas City, Missouri
  - Advanced Neurology Specialists (Benefis Healthcare Hospital), Great Falls, Montana
  - Washoe Comprehensive Stroke Center, Reno, Nevada
  - JFK Medical Center, Edison, New Jersey
  - Muhlenberg Regional Medical Center, Plainfield, New Jersey
  - Neurology Group of Bergen County (Valley Hospital), Ridgewood, New Jersey
  - University of New Mexico Hospital, Albuquerque, New Mexico
  - VA Medical Center, Albuquerque, New Mexico
  - Albany Medical Center, Albany, New York
  - Buffalo General Hospital, Buffalo, New York
  - North Shore University Hospital, Manhasset, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - Columbia Presbyterian Medical Center, New York, New York
  - Roosevelt Hospital, New York, New York
  - St. Luke's Hospital, New York, New York
  - Rochester General Hospital, Rochester, New York
  - Ellis Hospital, Schenectady, New York
  - Stony Brook Hospital, Stony Brook, New York
  - Forsyth Medical Center, Winston-Salem, North Carolina
  - Rowan Regional Medical Center, Winston-Salem, North Carolina
  - Akron General Medical Center, Akron, Ohio
  - Metrohealth Medical Center, Cleveland, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Medical College of Ohio, Toledo, Ohio
  - St. Elizabeth Health Center, Youngstown, Ohio
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Westmoreland Regional Hospital, Greensburg, Pennsylvania
  - Hershey Medical Center, Hershey, Pennsylvania
  - Albert Einstein Medical Center, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - University of Pennsylvania Medical Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center Stroke Institute, Pittsburgh, Pennsylvania
  - Crozer Chester Medical Center, Upland, Pennsylvania
  - Miriam Hospital, Providence, Rhode Island
  - Roper Hospital, Charleston, South Carolina
  - Chattanooga Neurology Associates (Erlanger Hospital), Chattanooga, Tennessee
  - Chattanooga Neurology Associates (Memorial Hospital), Chattanooga, Tennessee
  - St. Thomas Hospital, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas (Houston Medical Center), Houston, Texas
  - Neurological Research Center, Inc, Bennington, Vermont
  - Neurology Associates, Inc. (St. Mary's Hospital), Richmond, Virginia
  - Virginia Beach General Hospital, Virginia Beach, Virginia
  - Stevens Memorial Hospital, Edmonds, Washington
  - Providence St. Peter Hospital, Olympia, Washington
  - St. Luke's Medical Center, Milwaukee, Wisconsin
  - Theda Clark Medical Center, Neenah, Wisconsin
- Universitätsklinik allgemeines Krankenhaus der Stadt Wien, Vienna, Austria
- Dienst Neurologie UZ Gasthuisberg, Leuven, Belgium
- Canada (10):
  - Foothills Medical Centre, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - Penticton Regional Hospital, Penticton, British Columbia
  - Vancouver General Hospital, Vancouver, British Columbia
  - Royal Jubilee Hospital, Victoria, British Columbia
  - Victoria General Hospital, Victoria, British Columbia
  - Charles LeMoyne Hospital, Greenfield Park, Quebec
  - Notre-Dame Hospital, Montreal, Quebec
  - Pavillion St Joseph, Trois Rivers, Quebec
  - Royal University Hospital, Saskatoon, Saskatchewan
- Germany (12):
  - Universitätsklinikum Aachen, Neurologische Klinik, Aachen
  - Universität zu Köln klinik und poliklinik fur neurology, Cologne
  - University Essen, Essen
  - Neurologische Universitätsklinik, Freiburg im Breisgau
  - Universitätskrankenhaus Hamburg-Eppendorf Klinik für Neurologie, Hamburg-Eppendorf
  - Neurology Klinik Klinikum Hanover, Hanover
  - Friedrich-Schiller-University, Jena
  - Universitätsklinikum Leipzig, Leipzig
  - Universitätsklinik Mainz, Mainz
  - Neurologische Klinik Klinikum Rechts der Isar der TU Munchen, München
  - Neurologische Klinik Knappschafts - krankenhause, Recklinghausen
  - Neurologisch Psychiayrische Klinik, Weisbaden